CLINICAL TRIAL: NCT03992612
Title: Efficacy of Mindfulness-based Pain Management in Patients With Chronic Pain With and Without Fibromyalgia
Brief Title: Efficacy of Psychological Therapy in Chronic Pain and Fibromyalgia
Acronym: DOLORTRATPSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Karmele Salaberria, PhD. Lecturer in Psychology, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2018162
Record Dates: First submitted 2019-06-14; First posted 2019-06-20 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Fibromyalgia; Chronic Pain; Psychological Treatment; Effectiveness; MBPM
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): The patients received usual medical care.
  Interventions: Other: control group: usual medical care
- MBPM- Minfulness- Based Pain Management (Experimental): Psychological intervention with 8 group sessions ( 8 -10 subjects) with a duration of 2 and a half hours per session and a weekly periodicity (total hours 1080).
  It is centered on training on the awareness of physical, cognitive and emotional sensations, and the attentional processes to become an observer of one's own thoughts and emotions. With the aim to provide greater flexibility to manage pain
  Interventions: Behavioral: MBPM- Mindfulness-Based Pain Management

INTERVENTIONS:
Other: control group: usual medical care — The patients received usual medical care.
  Arms: control group
Behavioral: MBPM- Mindfulness-Based Pain Management — 8 group session of maindfulness-based treatment to management pain
  Arms: MBPM- Minfulness- Based Pain Management

SUMMARY:
Today, one of the most important challenges of the health system is the attitude towards chronic disorders. That implies changing from a health structure established for the treatment of acute diseases to a continued care system.

In this sense, the approach of chronic pain, of non-oncological origin, supposes an important care challenge, to which this project wishes to respond.

Chronic pain affects one of every Europeans (19%), and has a prevalence of 11% in Spain, being one of the most important causes of medical consultation and is associated with high personal, social and economic costs. For example, in 2017 it was calculated that it has an economic impact of between 1.7 and 2.1% of Spain's GDP.

Referred to the psychological consequences of the disease, it has been found that 42% of people who have chronic pain suffer insomnia, a 40% anxiety, and 24% depressive symptoms. Hence the importance of implementing evidence-based psychological treatments along with their treatment as usual The main objective is comparing the efficacy of mindfulness-based pain management (MBPM), together with the usual medical treatment, in patients diagnosed with chronic pain, with and without comorbid fibromyalgia.

Specific objectives are:

1. To study the sociodemographic and clinical profile of patients with chronic pain, with and without fibromyalgia.
2. Define the characteristics of patients who are in the different stages of the disease: stage 1 (less than two years since diagnosis); stage 2 (between 2 and 4 years); stage 3 (between 5 and 8 years), and stage 4 (more than 8 years).
3. Check the effectiveness of psychological therapies MBPM depending on the presence of fibromyalgia.
4. Check the effectiveness of the psychological treatment in function of the stage of the disease.

Method:

A quasi-experimental design of two groups will be used. Patients will be assigned to experimental group: 50 subjects will receive MBPM and control group 40 subjects, 3-months wait list, after which time they will also receive MBPM.

All the participants will be assessed in the baseline; at the end of the treatment; and in the 1, 3, 6 and 12 months follow-ups. Group 2 (waiting list) will be assessed in the baseline, and re-assessed before starting the treatment; at the end of the psychological therapy; and in the 1, 3, 6 and 12 months follow-ups.

DETAILED DESCRIPTION:
The objetive of this research are the study of efficacy in chronic pain and fybromyalgia of mindfulness therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be able to complete the assessment protocol
* Suffer from chronic non-oncological pain, lasting longer than 6 months
* Not being receiving psychological treatment
* Sign the informed consent

Exclusion Criteria:

* Present a cognitive impairment, such as a dementia
* Present a diagnosis of a psychotic disease, bipolar disease or additive disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Lattinen Index- IL | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  It is a scale with five items to assess variables associated with pain: frequency, intensity, disability, drugs usage and sleep problems. These are assessed by a Likert scale of 0 to 4, in order to explain the discomfort that pain generates. (Gonzalez-Escada, 2012)

SECONDARY OUTCOMES:
Change in the Fibromyalgia Impact Questionnaire- FIQ | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  its a 10 item scale that assesses the impact of the disease. The first item evaluates the interference of the disease in skills such as home care and work. The second item assesses how they felt last week; the third item values the days of last week that the disease prevented him from performing his usual tasks. Finally, the fourth item assesses the interference caused by pain and other items of the disease.
  It will only be completed by patients diagnosed with fibromyalgia. (Esteve et al., 2007)
Change in the Listado de Sintomas Breve- LSB-50 | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  it is composed of 50 items, which are rated on a Likert scale from 0 to 4, depending on the level of discomfort caused by each item to the subject. it includes two scales of validity, three general indices, clinical scales (psychoreactivity, hypersensitivity, obsession, anxiety, hostility, somatization, depression, and sleep disturbances) and a psychological risk index. (de Rivera & Abuin, 2012)
Change in the Short Form 12 Health Survey- SF-12 | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  It assesses a patient's health perception in 12 areas like physical function, physical role, body pain, general health, vitality, social function, emotional role, and mental health.
  It is completed with Likert type response options from 3 to 5 points.(Schmidt et al., 2012)
Change in Cuestionario de afrontamiento del dolor- CAD-R | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  It consists of 31 items related to the strategies that the patient performs when suffer pain. The strategies are valued from 1 (never use) to 5 (always use). The items are grouped into the following factors: religion, catharsis, distraction, information search, self-control, and self-affirmation. (Soriano & Monsaslve, 2002)
Change in Connor-Davison Resilience Scale- CDRISC | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  The CD-RISC scale assesses resilience. Consist in 25 items and the subject has to indicate what extent each of the statements has been true, in his case, during the last month on a scale ranging from 0 (not true at all) to 4 (almost always true). Fernández-Lansac & Soberón, 2014)
Change in Inventaire of negative thoughts in response to pain- INTRP | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  This questionnaire assesses the presence of negative thinking in response to pain. It consists of 21 items distributed in 5 factors: general negative thoughts, negative social thoughts, thoughts of disability, thoughts of lack of control, and thoughts of self-blame (Cano & Rodriguez, 2002)
Change Pain Catastrophizing Scale- PCS | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  The scale evaluates through 13 items the thoughts and feelings related to the experiences of pain. It is divided into three subscales, scored from 0 (never) to 4 (always), rumination, desperation, and magnification (Lami et al., 2013)
Change in Chronic Pain Acceptance Questionnaire- CPAQ | base line (week 0), end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  The scale evaluates strategies of the pain experience. It consists of 20 items, scored from 0 (never true) to 6 (always true), from which three scores are obtained: involvement in activities, openness to pain, and total punctuation.

OTHER OUTCOMES:
Client Satisfaction Questionnaire | end of treatment (week 12); and during maintenance phase (weeks 17, 29 and 41)
  This scale assesses clients satisfaction with the treatment through 8 items, using a Likert scale from 0 to 4. (Larsen et al., 1978)

CONTACTS AND LOCATIONS:
Overall Officials: Karmele Salaberria, PH.D, Principal Investigator — University of Basque Country
Locations (1):
- University of Basque Country, San Sebastián, Guipuzcoa, Spain